CLINICAL TRIAL: NCT02594462
Title: Use of Etonogestrel-releasing Contraceptive Implant in Women With Sickle Cell Disease
Brief Title: Contraception in Women With Sickle Cell Disease
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Sao Paulo (Other)
Collaborators: Escola Bahiana de Medicina e Saude Publica (Other)
Responsible Party: Principal Investigator, Milena Bastos Brito, MD, PhD, Milena Bastos Brito, University of Sao Paulo
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 458660
Record Dates: First submitted 2015-06-11; First posted 2015-11-03 (Estimated); Last update posted 2020-11-06 (Actual); Status verified 2020-11

CONDITIONS: Sickle Cell Disease
Keywords: contraception; Anemia, Sickle Cell
MeSH Terms: conditions — Anemia, Sickle Cell | interventions — etonogestrel

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- ENG-group (Other): Twenty-five women with homozygous sickle cell anemia (hemoglobin SS), aged between 18-40 years-old, who had at least one episode of sickle cell pain crisis in the last three months pre- enrollment; whom desire to use etonogestrel-releasing implant contraceptive without contraindications will be invited to inserted etonogestrel implant.
  Etonogestrel implant is a single implant progestogen-only, with 4 cm in length and 2 mm diameter containing 68 mg etonogestrel (3- ketodesogestrel), the active metabolite of desogestrel, involved in a ethylene vinyl acetate membrane (Huber, 1998), which is released continuously in bloodstream for three years. It will be inserted subdermal, on the inner face of non-dominant arm between the first and seventh day of the menstrual cycle.
  Interventions: Drug: etonogestrel-releasing implant contraceptive

INTERVENTIONS:
Drug: etonogestrel-releasing implant contraceptive — The etonogestrel implant will be inserted until the fifth day of the menstrual cycle . Anthropometric measurements will be performed , blood pressure measurement , application of pain questionnaire for the last three months, and collection of fasting blood in our clinic . After these measures , the ENG implant will be applied per researcher trained for such a procedure , following the recommendations outlined by the manufacturer. Women are instructed to return after 3, 6, 9, 12 months, fasting 8h , when they will be measured anthropometric measurements , blood collection, and delivery of pain questionnaires and standard of menstrual bleeding.
  Other Names: implanon

SUMMARY:
Sickle cell anemia is a homozygous genetic disease with high prevalence in Brazil. There are changes in conformation and physicochemical properties of red cells that generate varied clinical manifestations among which is chronic hemolytic anemia, cardiovascular diseases, fever, splenic sequestration and usually painful crises. Women with sickle cell anemia have high maternal-fetal and neonatal morbidity and mortality. During pregnancy, there is intensification of maternal anemia, episodes of painful crises; and also, more obstetric risks, such as pre-eclampsia, thromboembolism and hemorrhage. Thus, there is the need for adequate reproductive family planning for this population conducted mainly through hormonal contraception. The World Health Organization recommends that all contraceptive methods may be prescribed for people with sickle cell anemia women, being the progestogen-only contraceptive methods the most indicated due to no changes in venous or arterial thrombosis. Nevertheless, there is need for further scientific evidence as the best contraceptive choice among women with sickle cell anemia in relation to safety, adhesion and reduction of pain crises. The objective of this study is to evaluate the clinical effect through safety of etonogestrel-releasing contraceptive implant in women with sickle cell anemia during twelve months.

DETAILED DESCRIPTION:
There are 3,500 children born each year with sickle cell disease in Brazil. Almost three percent of Bahia population has sickle cell anemia, which is the most prevalent in Brazil (BRAGA, 2007).

Despite the high prevalence of sickle cell disease in our population, the best option Contraceptive for these women is still uncertain, based on low-quality studies (Haddad et al., 2012). Since this is a condition associated with numerous complications such as painful crises, splenic sequestration, marrow aplasia, among others, leads to frequent hospitalizations and high absenteeism rates. Women with sickle cell disease in reproductive age are exposed to non-planning pregnancies, which will cause high risk for maternal mortality (33%), and increased pictures of painful crises, and important maternal and newborn complications such as abortion, childbirth premature, thrombosis, among others (Andemariam, Browning, 2013). Therefore, there is a need to provide them with appropriate methods for effective reproductive planning.

Hormonal contraceptives with only progestogen, such as releasing implant etonogestrel (ENG), representing an option to reduce unwanted pregnancies, especially in patients at risk for venous thrombosis, such as patients with anemia sickle, because it doens´t interfere with the coagulation system (Conrad et al., 2004; Liedaagard etal., 2011). Thus, in addition to avoid an unwanted pregnancy, these methods have impact on reduction of maternal and fetal morbidity and mortality and neonatal known to be associated with pregnancies in women with sickle cell anemia (Santos et al., 2005).

The scientific literature is limited and scarce on the association between use of methods contraceptives in women with sickle cell disease and correlation with clinical complications such as seizures painful and anemia (Haddad et al., 2012).

The contraceptive implant etonogestrel is a reversibly progestogen-only contraceptive method, long lasting, highly effective, with high continuation rate. However, there is still no studies in women with sickle cell anemia in use thereof.

As it is a progestogen-only method, it does not increase the risk of thrombosis and may, as depot medroxyprogesterone acetate (Abood et al., 1997), reducing painful crises, with the advantage of high efficacy and long duration.

In this context, to increase adherence and whether a clinical benefit from use of the implant contraceptive releasing ENG, the contraceptive method more effectively isolated progestogen available in Brazil, in relation to painful crises and anemia among women with sickle cell disease, it is made of fundamental importance the development of a study in a city of high prevalence in Brazil.

ELIGIBILITY:
Inclusion Criteria:

1. Women with homozygous sickle cell anemia ( hemoglobin SS ) , who had at least one episode of sickle cell pain crisis in the last three months pre- enrollment.
2. Age between 18 and 40 years-old ;
3. Desire to use a long-term hormonal contraception
4. Agreed to participate in the study after reading and signing the informed consent form.

Exclusion Criteria:

1. Smoking, alcoholism or drug addiction ;
2. Obesity , defined as body mass index (BMI ) greater than or equal to 30 kg / m2 ;
3. contraindication to the use of isolated progestogen , according to WHO's eligibility criteria (WHO 2009)
4. Desire to maintain standard of cyclic menstrual bleeding ;
5. Allergy known local anesthetic ( lidocaine ) , once the implant is inserted after subdermal application of the local anesthetic

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 29 (Actual)
Dates: Start 2015-01; Primary Completion 2018-10 (Actual); Study Completion 2019-06 (Actual)

PRIMARY OUTCOMES:
Number of pain crises | 12 months
  Self reported of pain quantity on a diary.

SECONDARY OUTCOMES:
Clinical Safety as measured by hemoglobin, hepatic function | 12 months
  Immediately before the implant insertion, peripheral blood samples (20 mL) were collected Blood samples were collected to evaluate complete blood count (reticulocytes, hemoglobin, platelets and leukocytes), hepatic function (Alkaline phosphatase, gamma-glutaryl transferase, amino alanine transferase, aspartate amino transferase, total bilirubin and its fractions), before , 6 and 12 months after the implant insertion.
Pain Scores on the Visual Analog Scale | 12 months
  Pain intensity was measured by a visual scale, scored 0-10 (0=no pain until 10=worst pain) over each 3 months.

CONTACTS AND LOCATIONS:
Overall Officials: MILENA B BRITO, MD, PhD, Principal Investigator — University of Sao Paulo
Locations (2):
- Brazil (2):
  - Bahiana School of Medicne and Public Health, Salvador, Estado de Bahia
  - University of Sao Paulo, Ribeirão Preto, São Paulo

IPD SHARING:
Plan to Share IPD: No